CLINICAL TRIAL: NCT06726512
Title: Quantitative Margin Assessment Using High-resolution Positron Emission Tomography - Computed Tomograhy
Acronym: qMAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86142.042.24
Record Dates: First submitted 2024-10-16; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Oral Cancer; Osteosarcoma; Soft Tissue Sarcoma; Oral Squamous Cell Carcinoma (OSCC)
Keywords: margin assessment; image-guided surgery; PET-CT
MeSH Terms: conditions — Mouth Neoplasms; Osteosarcoma; Sarcoma; Squamous Cell Carcinoma of Head and Neck | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2 MBq 18F-FDG (Other): Subjects are intravenously administered with 2.0 MBq/kg 18F-FDG, standard tracer used to diagnose and stage the malignancy. After standard of care excision of the primary tumor, a high-resolution PET-CT imaging of the fresh surgical specimen will be performed.
  Interventions: Device: XEOS AURA 10

INTERVENTIONS:
Device: XEOS AURA 10 — Surgery is performed according to standard of care. Directly after surgery, the surgical specimen is taken outside the operation theatre in a dedicated imaging room at the Department of Nuclear Medicine where high-resolution PET-CT imaging of the surgical specimen is performed.
  Other Names: PET; PET/CT; High resolution PET/CT; Margin detection; Margin status

SUMMARY:
The primary endpoint is the assessment of the clinical value of a novel high-resolution mobile PET-CT scanner for intraoperative margin assessment in oral squamous cell carcinoma, soft tissue sarcoma and osteosarcoma surgery. The predicted margin status will be correlated with the margin status determined with histopathology.

DETAILED DESCRIPTION:
The ideal outcome in oncological surgery is resection of all tumor tissue with a margin of healthy tissue. However, positive surgical margins (PSMs) occur in up to 35% of the cases, depending on tumor type. The final margin status is only available five to seven days after surgery so that in case of a PSM, intensive adjuvant radiotherapy or chemotherapy is necessary. Despite adjuvant treatment, patients still have a significantly reduced overall survival. Therefore, the intraoperative identification of PSMs is paramount to enable surgical corrections and obtain a complete resection.

The investigators propose a dedicated intraoperative high-resolution PET-CT (positron emission tomography - computed tomography) imaging system for margin assessment of the excised specimen. The proposed specimen imaging system would combine the proven functional imaging capabilities of PET with the anatomical imaging info of CT, providing multi-modal information to determine whether tumor cells are present at the excision edges of the specimen. The tomographic images obtained can precisely demonstrate tumor extension along the x, y, and z axis, and the PET signal is not distorted by bone tissue. PET is the most sensitive medical imaging modality capable of detecting the picomolar concentrations of radiotracer, allowing to assess the presence of tumor cells within the specimen margins with high precision. Current standard PET-CT scanners have a spatial resolution between 3mm and 6mm, which is insufficient to accurately assess the excision margins of tumors. A specimen imaging system ideally should have a sub-millimeter resolution. The specimen PET system which will be used in this study is capable of this. The potential of intraoperative PET-CT has been shown in several tumor types, enabling the intraoperative identification of PSMs in prostatectomy and lumpectomy specimens.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patient is confirmed with oral squamous cell carcinoma, soft tissue sarcoma or osteosarcoma.
* Patient is indicated to undergo curative surgery of the primary tumor.
* Patient is estimated compliant for study participation by the investigator.
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Patient has previously received radiotherapy of the primary tumor region;
* Patient has participated in other clinical studies with radiation exposure of more than 1 mSv in the past 12 months;
* A blood glucose level over 200 mg/dL on the day of surgery.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to determine the margin detection rates of a novel high-resolution mobile PET-CT for intraoperative margin assessment in OSCC, STS, and OS surgery. | Postoperatively i.e. 7-10 working days
  Tumor positive and negative margin detection rates of the novel high-resolution mobile PET-CT scanner compared to standard of care pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Relevant research data on request
Supporting Information: Study Protocol, CSR
Time Frame: It will be available after the end date of the study. It will be available for 15 years after the study has ended.
Access Criteria: PI and other researchers on request. They are able to access the Study Protocol and the Clinical Study Report